CLINICAL TRIAL: NCT02978066
Title: Is Postspinal Hypotension a Sign of Impaired Cardiac Performance in the Elderly? An Observational Mechanistic Study
Brief Title: Postspinal Hypotension and Cardiac Performance in the Elderly
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sigridur Kalman, MD Professor, Karolinska Institutet
Other Study IDs: 2010-2042-31/1
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: ARTHROPLASTY, REPLACEMENT; ANESTHESIA
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Spinal anaesthesia

SUMMARY:
Patients, scheduled for elective arthroplasty were monitored with Lithium Dilution Cardiac Output monitor (LiDCOplus™) before and 45 minutes after spinal anesthesia. Hypotension was defined as systolic blood pressure ≤ 100 mmHg or ≥ 30% decrease from baseline. Associations between hypotension and the hemodynamic changes after preanaesthetic fluid loading and spinal anesthesia were analysed by logistic regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* hip or knee arthroplasty
* spinal anaesthesia
* age 65 years or more

Exclusion Criteria:

* weight <40kg
* concomitant lithium medication
* written informed consent not obtained
* research team unavailable

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years or older scheduled for hip or knee arthroplasty in spinal anaesthesia. Exclusion criteria were: (i) weight <40kg; (ii) concomitant lithium medication; (iv) informed consent not obtained; (v) research team unavailable
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Stroke volume in ml | 0-45 minutes after spinal anaesthesia
  the blood volume pumped by the heart at each stroke

SECONDARY OUTCOMES:
Arterial blood pressure mmHg and change from baseline | 0-45 minutes after spinal anaesthesia
  mmHg measured by arterial catheter

IPD SHARING:
Plan to Share IPD: No